CLINICAL TRIAL: NCT05593601
Title: Decolonization of Carbapenem-resistant Enterobacterales (CRE) in Patients With Faecal Carriage of CRE With Neomycin
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SI-CEU-02-2022
Record Dates: First submitted 2022-10-17; First posted 2022-10-25 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Colonization, Asymptomatic
Keywords: Neomycin; CRE; carbapenem-resistant Enterobacterales
MeSH Terms: conditions — Asymptomatic Infections | interventions — Neomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neomycin (Active Comparator): Patients enrolled in this arm will receive Neomycin.
  Interventions: Drug: Neomycin
- Non neomycin (No Intervention): Patients enrolled in this arm will not receive any interventions.

INTERVENTIONS:
Drug: Neomycin — Neomycin (350 mg/tablet) 1.4 g three times a day (4.2 g per day) for 5 days
  Other Names: Neomycin Sulfate
  Arms: Neomycin

SUMMARY:
Rates of antimicrobial resistance are increasing worldwide. There is increasing evidence that physiological gut microbiota is a large reservoir of antibiotic-resistance genes. Healthy gut microbiota is known to prevent the colonization of the gastrointestinal tract by pathogens, the so-called mechanism of colonization resistance, but this protective mechanism can be altered by therapies that impair gut microbiota, including antibiotics with consequent colonization of gut pathogens, including carbapenem-resistant Enterobacterales (CRE). CRE carriers represent an epidemiological threat to other hospitalized patients and to the whole community, but are also at risk of developing clinical consequences of this colonization, including bloodstream infections from these pathogens. Neomycin has shown high efficacy in the eradication of CRE invitro. Neomycin has also been approved to treat hepatic coma by eradicating bacterial in gastrointestinal tract. Therefore, this evidence suggests that this procedure could be useful in eradicating CRE.

However, current evidence is mostly limited.

The aim of this study is to investigate the efficacy of Neomycin, compared with no intervention in eradicating gut colonization from CRE.

DETAILED DESCRIPTION:
The investigators will randomize patients colonized by CRE (diagnosed by rectal swab) to Neomycin by stratified randomization according to type of CRE species (E.coli or non-E.coli). Then, patients will be followed up, rectal swabs will be repeated, and stool samples for culture and will be collected, up to 14 days after Neomycin.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged >18 years
* Hospitalized in medical wards
* Presence of CRE in stool/rectal swab without symptom from active surveillance of CRE
* Sign informed consent to participate the study

Exclusion Criteria:

* CRE infected patients
* Receiving anti-CRE antibiotics
* Known allergy to neomycin or other aminoglycosides
* Receiving Cidofovir, Colistin methate sodium, foscarnet , furosemide, digoxin
* eGFR (estimated Glomerular Filtration Rate) < 30 ml/min/1.73 m2
* Had gastro-intestinal tract diseases
* Pregnancy or breast-feeding

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-24 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with microbiological eradication at 2 weeks after neomycin administration | 2 weeks
  Microbiological eradication is defined as the disappearance of CRE in hospitalized patients' faces at 2 weeks after neomycin administration

SECONDARY OUTCOMES:
Incidence of ์Neomycin toxicity (safety) | 2 weeks
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0
Incidence of ์carbapenemases in isolated CRE | 2 weeks
  Number of carbapenemases in isolated CRE
Number of CRE isolates susceptible to neomycin at 2 weeks after neomycin administration | 2 weeks
  Number of CRE isolates are susceptible to neomycin at 2 weeks after neomycin administration according to the Clinical and Laboratory Standards Institute (CLSI) guideline.
Number of CRE isolates susceptible to amikacin at 2 weeks after neomycin administration | 2 weeks
  Number of CRE isolates are susceptible to amikacin after at 2 weeks after neomycin administration according to the Clinical and Laboratory Standards Institute (CLSI) guideline.
Number of CRE isolates susceptible to gentamicin at 2 weeks after neomycin administration | 2 weeks
  Number of CRE isolates are susceptible to gentamicin at 2 weeks after neomycin administration according to the Clinical and Laboratory Standards Institute (CLSI) guideline.

CONTACTS AND LOCATIONS:
Overall Officials: Adhiratha Boonyasiri, MD, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hu Y, Liu L, Zhang X, Feng Y, Zong Z. In Vitro Activity of Neomycin, Streptomycin, Paromomycin and Apramycin against Carbapenem-Resistant Enterobacteriaceae Clinical Strains. Front Microbiol. 2017 Nov 17;8:2275. doi: 10.3389/fmicb.2017.02275. eCollection 2017. PMID 29250040
- [Background] Park SY, Lee JS, Oh J, Lee SH, Jung J. Effectiveness of selective digestive decolonization therapy using oral gentamicin for eradication of carbapenem-resistant Enterobacteriaceae carriage. Infect Control Hosp Epidemiol. 2022 Nov;43(11):1580-1585. doi: 10.1017/ice.2021.492. Epub 2022 Feb 9. PMID 35135653